CLINICAL TRIAL: NCT03355417
Title: A Multiple Baseline Design Study to Investigate the Effectiveness of OT-SI Using an Intensive Intervention Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20012008
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Motor Coordination or Function; Developmental Disorder
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: This study will use a non-concurrent multiple baseline design (MBD) where subjects will serve as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OT-SI (Experimental): Occupational therapy using a sensory integration approach
  Interventions: Other: OT-SI

INTERVENTIONS:
Other: OT-SI — Occupational therapy using a sensory integration approach (OT-SI) 3x per week for 10 weeks. A typical session will be 1 hour (total of 3 hours per week).

SUMMARY:
The investigators hypothesize that children completing 30 sessions of occupational therapy using a sensory integration approach (OT-SI) will demonstrate positive changes in outcome measures related to motor coordination, functional performance and sensory processing (changes pre-post test).

ELIGIBILITY:
Inclusion Criteria:

* Have a medical diagnosis of "lack of coordination" or "other coordination impairment"
* Children and caregivers able to communicate verbally in English
* Sensory processing impairments as determined by scores in the SPM-H form (screening). Scores must fall in the "definite dysfunction" range in one of three categories (Body Awareness, Balance & Motion, or Planning & Ideas), OR fall in the "some problems" range in 2/3 areas.

Exclusion Criteria:

* Diagnosed with autism spectrum disorder or other significant psychological impairment (e.g. bipolar disorder)
* Receiving occupational therapy services at CHoR or another therapy site for more than 3 months
* Significant motor impairment (e.g., cerebral palsy)
* Significant language impairment (e.g., non-verbal, or aphasia)

Ages: 59 Months to 107 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Change in motor coordination: Jumping Jacks | Baseline to 10 weeks
  Amount of correct jumps in specified time frame (10 seconds)
Change in motor coordination: Finger to Nose Touching | Baseline to 10 weeks
  Amount of correct touches in specified time frame (10 seconds)
Change in motor coordination: Single Leg Stance Balance | Baseline to 10 weeks
  Time held in seconds

SECONDARY OUTCOMES:
Change in Sensory Processing Measure-Home Form | Baseline to 10 weeks
  A standardized set of questionnaires used for rating a child's sensory processing issues, motor planning (praxis), and social participation.
Change in Bruinincks-Oseretsky Test of Motor Proficiency (BOT-2) Short-Form | Baseline to 10 weeks
  A standardized assessment that uses goal-directed motor activities to measure a wide array of gross and fine motor skills in individuals 4-21 years old.
Change in Goal Attainment Scaling | Baseline to 10 weeks
  Goal Attainment Scaling (GAS) is a way to develop individual goals for a patient that can be measured over the course of intervention using a standardized scale. Goals are rated on a 5-point scale and criteria for each level is established prior to starting treatment. While each patient has individual goals that are meaningful to him/her and his/her family, the outcome measurement scale is standardized so that it can be used for statistical analysis with other patients' goals. The expected level of outcome is established at initial goal setting, and 0 is used to rate an outcome where a patient achieves the expected level. If patient achieves a better than expected outcome, the score can be +1 (somewhat better) or +2 (much better). If patient achieves a worse outcome than expected, the score can be -1 (somewhat worse) or -2 (much worse). GAS goals are identified during semi-structured interview with patient and/or caregivers, and 3-4 goals are set and weighted by importance.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Reynolds, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States